CLINICAL TRIAL: NCT04123938
Title: A Pilot Study to Examine the Effect of Pea Protein on Limiting the Loss of Muscle Mass During Weight Loss
Brief Title: Pea Protein and Muscle Mass During Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Peter Zahradka, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS22196
Record Dates: First submitted 2019-09-26; First posted 2019-10-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Pea Proteins; Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pea Protein (Experimental): Participants will consume pea protein (0.35 grams protein/kg body weight/day) as a powder incorporated into foods or beverages at least twice per day for 12 weeks.
  Interventions: Other: Pea Protein
- Whey Protein (Active Comparator): Participants will consume whey protein (0.35 grams protein/kg body weight/day) as a powder incorporated into foods or beverages at least twice per day for 12 weeks.
  Interventions: Other: Whey Protein
- Maltodextrin (Placebo Comparator): Participants will consume maltodextrin (isocaloric non-protein comparator) as a powder incorporated into foods or beverages at least twice per day for 12 weeks.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Pea Protein — Soluble pea protein
  Other Names: NUTRALYS S85
  Arms: Pea Protein
Other: Whey Protein — Whey protein concentrate
  Other Names: Whey Protein Concentrate 80 Instant Kosher
  Arms: Whey Protein
Other: Maltodextrin — Non-protein isocaloric comparator
  Other Names: GLUCIDEX 19
  Arms: Maltodextrin

SUMMARY:
A pilot study comparing the effects of pea protein versus whey protein on the preservation of muscle mass and functionality in individuals undertaking a weight loss regimen.

DETAILED DESCRIPTION:
A single site, double-blind, randomized clinical trial designed to compare the effects of pea protein or whey protein or maltodextrin supplementation on muscle mass and functionality in males and females with obesity undertaking a weight loss regimen. Eligible participants will be randomized to one of the three groups (pea protein, whey protein, maltodextrin) and will be asked to attend 3 in-person clinic visits (0, 6, and 12 weeks) for blood and urine collection and assessments of muscle mass and muscle function. A separate visit for screening and for a fasting blood sample, as well as a Pre-Study visit and a meeting with a registered dietitian, will be required.

ELIGIBILITY:
Inclusion Criteria:

1. Male, or non-pregnant, non-lactating female, 30 to 50 years of age;
2. BMI >30 and body weight does not exceed the capacity of the DEXA (350 lbs);
3. Fat mass >23% for males and >32% for females (determined at the screening visit via bioelectrical impedance);
4. Willing to maintain a stable level of activity while participating in the study;
5. Plasma creatinine ≤265 µmol/L;
6. Plasma LDL-cholesterol <5 mmol/L;
7. Aspartate aminotransferase <160 U/L, and alanine aminotransferase <150 U/L;
8. Glycated hemoglobin <6.5%;
9. Blood pressure <160 mmHg systolic and <100 mmHg diastolic;
10. Stable regime if taking vitamin and mineral/dietary/herbal supplements for the past 1 month and while participating in the study;
11. Not taking protein supplements for the past month and willing to continue doing so for the duration of the study;
12. Has not donated blood or blood products (e.g. platelets) during the past 2 months and willing to continue doing so while participating in the study;
13. Female participants of child-bearing potential must agree to use a highly effective method of contraception throughout the study;
14. Not participating in another dietary intervention trial for the past month and willing to not start another dietary intervention trial or weight loss program for the duration of this study;
15. Willing to comply with the protocol requirements and procedures;
16. Willing to provide informed consent.

Exclusion Criteria:

1. Has experienced a cardiovascular event (e.g. heart attack, stroke) or had a surgical procedure for cardiovascular disease (e.g. bypass, stent), presence of diabetes, chronic renal disease, liver disease (with exception of fatty liver), rheumatoid arthritis, immune disorder or disease (e.g. multiple sclerosis, leukemia), cancer in the previous 5 years, neurological disorders, gastrointestinal disorders or gastrointestinal surgery or bariatric surgery, or liposuction;
2. Taking medications for blood glucose management;
3. Taking medications or natural health products/supplements associated with weight gain or weight loss (e.g. prednisone, certain cold medications);
4. Body weight that has not been stable (± 5%) over the past 3 months;
5. History of gastrointestinal reactions or allergies to peas, pea protein, whey protein or maltodextrin, or to one or more ingredients in the beverages and foods that will be provided which significantly limits the number of items that can be used for delivery of the protein powders or maltodextrin;
6. Current (within the past 30 days) bacterial, viral or fungal infection;
7. Uncontrolled hypothyroidism;
8. Uncontrolled blood pressure;
9. Bleeding disorder;
10. Any acute medical condition or surgical intervention within the past 3 months;
11. Cigarette/cigar smoking or use of tobacco products within the last 12 months or during participation in the study;
12. Consumption of >10 alcoholic beverages per week or >2 alcoholic beverages per day within the last 3 months or while participating in the study;
13. Drug and/or alcohol abuse;
14. Psychological disorder(s);
15. Unable to obtain blood sample at the screening or week 0 visits.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | Baseline and 12 weeks
  Muscle mass will be assessed by dual x-ray absorptiometry
Change in muscle function (hand grip) | Baseline and 12 weeks
  A dynamometer will be used to measure hand grip strength
Change in muscle function (gait test) | Baseline and 12 weeks
  A gait test will be performed

SECONDARY OUTCOMES:
Change in fat mass | Baseline and 12 weeks
  Fat mass will be measured by dual x-ray absorptiometry
Change in body weight and body mass index | Baseline and 12 weeks
  Body weight will be measured and used for calculation of body mass index
Change in waist and waist to height ratio | Baseline and 12 weeks
  Waist circumferences will be measured and used for calculation of waist to height ratio
Change in resting energy expenditure | Baseline and 12 weeks
  Resting energy expenditure will be measured by metabolic cart
Change in C-reactive protein | Baseline and 12 weeks
  A fasting venous blood sample will be analyzed for C-reactive protein to assess inflammatory status
Change in homeostatic model for insulin resistance (HOMA-IR) | Baseline and 12 weeks
  A fasting venous blood sample will be analyzed for insulin and glucose to calculate HOMA-IR using the formula fasting insulin x fasting glucose / 405
Change in glycated hemoglobin | Baseline and 12 weeks
  A fasting venous blood sample will be analyzed for glycated hemoglobin
Change in blood lipid profile | Baseline and 12 weeks
  A fasting venous blood sample will be analyzed for total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides as the blood lipid profile
Change in kidney function (based on profile of circulating markers) | Baseline and 12 weeks
  A fasting venous blood sample will be analyzed for blood urea nitrogen and serum creatinine to obtain a profile of circulating markers for assessing kidney function
Change in kidney function (based on profile of urinary markers) | Baseline and 12 weeks
  A spot urine sample will be analyzed for urine albumin, creatinine and urea to obtain a profile of urinary markers for assessing kidney function
Change in liver function (based on profile of circulating markers) | Baseline and 12 weeks
  A fasting venous blood sample will be analyzed for plasma alanine aminotransferase and aspartate aminotransferase to obtain a profile of circulating markers for assessing liver function
Change in systolic and diastolic blood pressure | Baseline and 12 weeks
  Systolic and diastolic blood pressure will be measured
Changes in blood vessel function | Baseline and 12 weeks
  Pulse wave velocity measurements will obtained for assessment of arterial stiffness, an indicator of blood vessel function
24 h activity patterns over time | Up to 12 weeks
  Participants will wear a Fitbit to monitor 24 hour activity patterns
Food intake over time | Up to 12 weeks
  Participants will complete 3-Day Food Records at 3 week intervals for analysis of nutrient intake

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zahradka, PhD, Principal Investigator — St. Boniface Hospital Albrechtsen Research Centre
Locations (1):
- I.H Asper Clinical Research Institute, St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No